CLINICAL TRIAL: NCT05969405
Title: Comparison of Prognosis in Endometrial Cancer Treated With Different Surgical Methods: Laparoscopy, Robotic-assisted Laparoscopy and Laparotomy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Sheng-Mou Hsiao, Chief, Department of Obstetrics & Gynecology, Far Eastern Memorial Hospital
Other Study IDs: 112002-E
Record Dates: First submitted 2023-07-23; First posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Laparoscopy: Laparoscopic staging group
  Interventions: Procedure: Laparoscopic staging
- Robotic: Robotic staing group
  Interventions: Procedure: Robotic staging
- Laparotomic: Laparotomic group
  Interventions: Procedure: Laparotomic staging

INTERVENTIONS:
Procedure: Laparoscopic staging — Laparoscopic staging
  Groups: Laparoscopy
Procedure: Robotic staging — Robotic staging
  Groups: Robotic
Procedure: Laparotomic staging — Laparotomic staging
  Groups: Laparotomic

SUMMARY:
Objective：To compare the clinical outcomes of endometrial cancer patients who received surgerical treatments: Comparisons of robotic-assisted laparoscopic, laparoscopic and laparotomic methods

DETAILED DESCRIPTION:
We will review the medical records of clinically uterine-confined endometrial cancer women who received robotic-assisted laparoscopic, laparoscopic or laparotomic methods; and compare their outcomes.

ELIGIBILITY:
Inclusion Criteria:

* womwn who received endometrial cancer surgical from January 01, 2008 to November 30, 2022 were be reviewed.

Exclusion Criteria:

* Endometrial cancer patients did not undergo surgery.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women with endometrial cancer who were treated in Far Eastern Memorial Hospital from January 01, 2008 to November 30, 2022 were be reviewed.
Study Population: endometrial cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-07-07 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 5 years
  Overall survival

SECONDARY OUTCOMES:
Progression free survival | 5 years
  Progression free survival
length of hospital stay | 2 weeks
  length of hospital stay
surgical time | 1 day
  surgical time
Estimate blood loss | 1 day
  Estimate blood loss
lymph node number | 1 day
  dissected lymph node number

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstetrics and Gynecology, Far Eastern Memorial Hospital, Banqiao District, New Taipei, Taiwan